CLINICAL TRIAL: NCT04180566
Title: Does Weekly Antepartum Testing in Women With BMI 30-40 Improve Neonatal Outcomes: A Randomized Controlled Trial
Brief Title: Weekly Antepartum Testing in Women With BMI 30-40 and Neonatal Outcomes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AAAS5275
Record Dates: First submitted 2019-11-26; First posted 2019-11-27 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Obesity Complicating Childbirth
Keywords: Pregnant; Pregnancy; Ultrasound; Antepartum testing; Neonatal outcome; Antenatal complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weekly antenatal testing (Other): Women with BMI 30-40 between 20 and 34.6 weeks of gestation will receive weekly antenatal testing (biophysical profile) starting at 34 weeks as well as growth ultrasound every 4 weeks.
  Interventions: Other: Antenatal Testing (biophysical profile)
- Growth ultrasound examination every 4 weeks (Other): Women with BMI 30-40 between 20 and 34.6 weeks of gestation will receive ultrasound examination (growth ultrasound) every 4 weeks starting at 34 weeks.
  Interventions: Other: Ultrasound Examination

INTERVENTIONS:
Other: Ultrasound Examination — Includes a regular growth ultrasound examination.
  Arms: Growth ultrasound examination every 4 weeks
Other: Antenatal Testing (biophysical profile) — Includes weekly ultrasounds with a biophysical profile, which measures fetal tone, fetal movements, fetal breathing and amount of amniotic fluid (water around baby).
  Arms: Weekly antenatal testing

SUMMARY:
The purpose of study is to evaluate whether weekly antenatal testing in pregnant women with body mass index (BMI) 30-40 in the third trimester is associated with earlier delivery when compared to growth ultrasounds every 4 weeks. The investigators will also assess the differences in maternal and neonatal outcomes between the groups.

DETAILED DESCRIPTION:
Over the last decade, the prevalence of obesity has dramatically increased in women in reproductive age. It is well known that obesity has been associated with increased risk of antenatal complications, maternal and perinatal morbidity, including higher risk of stillbirth. Studies including obese women without other antepartum comorbidities have shown that up to 11% of pregnancies are complicated with fluid and fetal growth abnormalities. According to American College of Obstetricians and Gynecologists (ACOG) guidelines, antepartum surveillance has not been proven to improve pregnancy outcomes in such cases and no specific recommendations for antepartum surveillance in obese women have been established.

ELIGIBILITY:
Inclusion Criteria:

* Women at or over 18 years of age
* Singleton pregnancy with no major fetal anomalies
* Pregnancies and gestational age will be well dated
* Obese with BMI 30-40kg/m2

Exclusion Criteria:

* Women with any complications at time of randomization that would require antenatal testing in the third trimester as per ACOG guidelines including: hypertension, systemic lupus erythematosus, chronic renal disease, antiphospholipid syndromes, hyperthyroidism poorly controlled, hemoglobinopathies, cyanotic heart disease, gestational hypertension, pre-eclampsia, gestational diabetes medication controlled, oligohydramnios, intrauterine growth restriction before randomization, isoimmunization, history of fetal demise
* Women with indication for weekly testing as per local protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
Average gestational age at delivery of participating women's babies | At time of delivery
  This is to measure the number of weeks that the baby has been in the uterus. It is measured from the first day of the woman's last menstrual cycle to the date of delivery. A normal pregnancy can range from 38 to 42 weeks. A significant delay in gestational age of delivery would be > 7 days out of this range.

SECONDARY OUTCOMES:
Average birth weight of participating women's babies | At time of delivery
  This is to measure the body weight of a baby at birth. The average baby weighs about 7.5 pounds - though the range of normal is between 5.8 and 10 pounds.
Number of participating women who experienced composite maternal morbidity | At time of delivery
  Composite maternal morbidity is defined as any of the following: chorioamnionitis, endometritis, cesarean section in labor, wound infection, transfusion, hemorrhage, deep venous thrombosis or pulmonary embolism, admission to ICU or death.
Number of participating women whose babies experienced composite neonatal morbidity | At time of delivery
  Composite neonatal morbidity is defined as any of the following: stillbirth after randomization, neonatal death within 28 days from birth, respiratory distress syndrome, Transient tachypnea of the newborn, hypoglycemia, sepsis, seizures, necrotizing enterocolitis, hypoxic ischemic encephalopathy, cardiopulmonary resuscitation or ventilator support within 24 h of birth, arterial blood pH<7, 5 min Apgar score <3, ICU admission, prolonged hospitalization (5 days or longer).
Number of participating women whose babies experienced composite of abnormalities of fluid volume and growth | At time of delivery
  A composite of abnormalities of fluid volume and growth is defined as any of the following: oligohydramnios (AFI<5 or maximum vertical pocket (MVP) < 2) or polyhydramnios (AFI>24 or MVP>8); fetal growth restriction (EFW<10% or AC<5%) ; or large for gestational age (EFW>90%), macrosomia (EFW>4,000 grams).

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Gyamfi-Bannerman, MD, MSc, Principal Investigator — Professor of Obstetrics/Gyn, Columbia University; Maria Andrikopoulou, MD, PhD, Study Chair — Postdoctoral Clinical Fellow in the Department of Obstetrics
Locations (1):
- Columbia Univeristy Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided